CLINICAL TRIAL: NCT05015634
Title: Remote Acute Assessment of Patients With High Cardiovascular Risk Post-Acute Coronary Syndrome
Brief Title: Telemedicine in High-Risk Cardiovascular Patients Post-ACS
Acronym: TELE-ACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: King Khalid University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21HH7034
Record Dates: First submitted 2021-08-11; First posted 2021-08-20 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases; Acute Coronary Syndrome
Keywords: Myocardial infarction; Acute coronary syndrome; Telemedicine; Heart Attack
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: A total of 338 patients will be randomised 1:1 to the 2 trial arms over 9 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Arm (Active Comparator): Patients will be discharged from the hospital with the telemedicine package. If the patient develops possible cardiac symptoms and seeks medical attention, the data provided by the telemedicine package will be acted upon, as appropriate, by the trial cardiology team. With remote follow up over the phone at 3, 6 and 9 months.
  Interventions: Other: Active Arm
- Control Arm (Placebo Comparator): Standard routine clinical care will be carried out, with remote follow up over the phone at 3, 6 and 9 months.
  Interventions: Other: Control Arm

INTERVENTIONS:
Other: Active Arm — Patient develops possible cardiac symptoms, takes an ECG, BP and oxygen saturation as per their training. Patient will receive a phone call by the trial cardiologist who will have access to a high-quality ECG trace, as well as blood pressure and oxygen saturations, and coupled with the clinical history, can decide on the most appropriate course of further management. With remote follow up over the phone at 3, 6 and 9 months.
  Arms: Active Arm
Other: Control Arm — Standard routine clinical care will be carried out, with remote follow up over the phone at 3, 6 and 9 months.
  Arms: Control Arm

SUMMARY:
This is a non-CTIMP randomised controlled trial looking at the utilisation of telemedicine devices to provide remote, clinically necessary, diagnostic information, without the need for hospital attendance that patients will take home with them following admission to hospital with a heart attack.

DETAILED DESCRIPTION:
Following hospital admission with a heart attack, telemedicine equipment can provide patients with remote, clinically necessary diagnostic information without the need for hospital attendance, which they can take home when they discharge from the hospital. In this project, patients known to be at high risk of ACS are equipped and empowered to seek urgent medical attention without visiting the hospital, if they experience symptoms, and to determine whether or not to seek emergency treatment, with an immediate remote specialist consultation, as assessed by validated technology.

Those enrolled in the intervention group will be offered telemedicine packages upon discharge from the hospital. Those enrolled in the active arm will have their telemedicine package provided to the trial team when they conduct an ECG and seek medical attention. In contrast, in the control group, routine clinical care will be provided, as well as follow up by phone over 9 months.

ELIGIBILITY:
Inclusion Criteria:

* 1 ACS Patients diagnosed with elevated hs-cTnI I who have undergone coronary intervention for NSTEMI or STEMI or unstable angina.
* 2 In addition, the participant should have at least one additional cardiovascular risk factor:

  * Current or ex-Tobacco Use
  * Hypertension
  * Diabetes
  * Hypercholesterolaemia.
  * Male aged > 50 years.
* 3 Access to a smartphone or smart device.

Exclusion Criteria:

* 1 The inability to apply/use the telemonitoring equipmentt
* 2 Life expectancy of 9 months or less.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
All hospital readmission rates | 6 months
  At 6 months of follow up, compare formal admissions and not emergency room visits in intervention to control groups.

SECONDARY OUTCOMES:
Length of stay | 9 months
  Length of stay at 3, 6, and 9 months will be compared in both study groups.
All-cause mortality, morbidity, and MACE. | 9 months
  At 9 months of follow up, compare all-cause mortality, morbidity, and MACE.
Medical intervention | 9 months
  Compare Medical intervention for for acute coronary syndromes or heart failure, including coronary angiography/ angioplasty, injectable therapy or oxygen therapy for both study groups when readmission to hospital.
Emergency Department visits | 9 months
  Any emergency department visits not requiring admission or further intervention will be compared in both study groups at 9 months of follow up.
9 months readmission rates | 9 months
  The readmission rates for 9 months will be compared in both study groups.
Patient-reported quality of life | 9 months
  Patients in both study groups will fill out a quality of life questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi Y Khamis, MB ChB PhD FRCP, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Once the study is complete and analysed, whilst individual patient results will not be disclosed, the overall research findings may be submitted for publication in a scientific journal and presented at scientific conferences following the completion of the study. A summary of the research findings will be uploaded onto the Imperial College London website. All data will be anonymised and kept confidential.

REFERENCES:
- [Background] Kwok CS, Wong CW, Shufflebotham H, Brindley L, Fatima T, Shufflebotham A, Barker D, Pawala A, Heatlie G, Mamas MA. Early Readmissions After Acute Myocardial Infarction. Am J Cardiol. 2017 Sep 1;120(5):723-728. doi: 10.1016/j.amjcard.2017.05.049. Epub 2017 Jun 15. PMID 28728745
- [Background] Wang H, Zhao T, Wei X, Lu H, Lin X. The prevalence of 30-day readmission after acute myocardial infarction: A systematic review and meta-analysis. Clin Cardiol. 2019 Oct;42(10):889-898. doi: 10.1002/clc.23238. Epub 2019 Aug 12. PMID 31407368
- [Background] Southern DA, Ngo J, Martin BJ, Galbraith PD, Knudtson ML, Ghali WA, James MT, Wilton SB. Characterizing types of readmission after acute coronary syndrome hospitalization: implications for quality reporting. J Am Heart Assoc. 2014 Sep 18;3(5):e001046. doi: 10.1161/JAHA.114.001046. PMID 25237046
- [Background] Dreyer RP, Dharmarajan K, Kennedy KF, Jones PG, Vaccarino V, Murugiah K, Nuti SV, Smolderen KG, Buchanan DM, Spertus JA, Krumholz HM. Sex Differences in 1-Year All-Cause Rehospitalization in Patients After Acute Myocardial Infarction: A Prospective Observational Study. Circulation. 2017 Feb 7;135(6):521-531. doi: 10.1161/CIRCULATIONAHA.116.024993. PMID 28153989
- [Background] Khera R, Wang Y, Bernheim SM, Lin Z, Krumholz HM. Post-discharge acute care and outcomes following readmission reduction initiatives: national retrospective cohort study of Medicare beneficiaries in the United States. BMJ. 2020 Jan 15;368:l6831. doi: 10.1136/bmj.l6831. PMID 31941686
- [Background] Ben-Assa E, Shacham Y, Golovner M, Malov N, Leshem-Rubinow E, Zatelman A, Oren Shamir A, Rogowski O, Roth A. Is telemedicine an answer to reducing 30-day readmission rates post-acute myocardial infarction? Telemed J E Health. 2014 Sep;20(9):816-21. doi: 10.1089/tmj.2013.0346. Epub 2014 Jul 21. PMID 25046174
- [Background] Garcia S, Albaghdadi MS, Meraj PM, Schmidt C, Garberich R, Jaffer FA, Dixon S, Rade JJ, Tannenbaum M, Chambers J, Huang PP, Henry TD. Reduction in ST-Segment Elevation Cardiac Catheterization Laboratory Activations in the United States During COVID-19 Pandemic. J Am Coll Cardiol. 2020 Jun 9;75(22):2871-2872. doi: 10.1016/j.jacc.2020.04.011. Epub 2020 Apr 10. No abstract available. PMID 32283124
- [Background] Marijon E, Karam N, Jost D, Perrot D, Frattini B, Derkenne C, Sharifzadehgan A, Waldmann V, Beganton F, Narayanan K, Lafont A, Bougouin W, Jouven X. Out-of-hospital cardiac arrest during the COVID-19 pandemic in Paris, France: a population-based, observational study. Lancet Public Health. 2020 Aug;5(8):e437-e443. doi: 10.1016/S2468-2667(20)30117-1. Epub 2020 May 27. PMID 32473113
- [Derived] Alshahrani NS, Hartley A, Howard J, Hajhosseiny R, Khawaja S, Seligman H, Akbari T, Alharbi BA, Bassett P, Al-Lamee R, Francis D, Kaura A, Kelshiker MA, Peters NS, Khamis R. Randomized Trial of Remote Assessment of Patients After an Acute Coronary Syndrome. J Am Coll Cardiol. 2024 Jun 11;83(23):2250-2259. doi: 10.1016/j.jacc.2024.03.398. Epub 2024 Apr 6. PMID 38588928